CLINICAL TRIAL: NCT05375149
Title: Exhaled Breath Particles as a Clinical Indicator for Acute and Chronic Rejection After Lung Transplantation
Brief Title: Exhaled Breath Particles in Lung Transplantation
Status: Recruiting | Type: Observational
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LTxPEx
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-02

CONDITIONS: Lung Transplant Rejection; Primary Graft Dysfunction; Chronic Rejection of Lung Transplant
Keywords: Exhaled Breath Particles; PExA; Lung transplantation; Primary Graft Dysfunction; Chronic Lug Allograft Dysfunction
MeSH Terms: conditions — Primary Graft Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Exhaled breath particles (EBP), blood samples, bronchoalveolar lavage fluid (BAL), biopsies of lung tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LTx rejection: Lung transplanted patients with acute or chronic rejection
- LTx non-rejection: Lung transplanted patients without any form of rejection

SUMMARY:
Lung transplantation (LTx) is the only effective treatment for patients with end stage lung disease. Of the major organs transplanted, survival following LTx is the lowest with a mean of 5 years. Despite improvements, primary graft dysfunction (PGD) remains the leading cause of early mortality and contributes to the development of chronic lung allograft dysfunction (CLAD) that remains the leading cause of late mortality. Earlier detection of rejection after LTx is of substantial importance as it would improve the possibilities of treatment and could increase survival.

The investigators have shown in previous work that exhaled breath particles (EBP) reflect the composition of respiratory tract lining fluid (RTLF). EBP and particle flow rate (PFR) can be used as non-invasive methods for early detection and monitoring of airway diseases such as acute respiratory distress syndrome (ARDS). It has also been shown that the particle flow prolife after lung transplantation differs between patients who develop PGD and those who do not and that the composition of EBP differs between patients with and without bronchiolitis obliterans syndrome (BOS), an obstructive form of CLAD.

Samples of EBP and measurements of PFR will be collected from lung transplanted patients. Membranes with EBP will be saved for molecular analysis. The investigators aim to identify potential particle flow patterns and biomarkers for earlier detection of rejection after lung transplantation.

DETAILED DESCRIPTION:
Samples of EBP and measurement of PFR will be done on patients undergoing lung transplantation at Skåne University Hospital (SUS) Lund. Measurements of EBP and PFR and collection of blood will be done repeatedly postoperatively when the patient is still in the hospital, at three months post-transplantation, at six months post-transplantation, at 12 months post-transplantation and annually after that. An additional preoperative blood sample will also be obtained. Furthermore, the investigators will collect bronchoalveolar lavage fluid (BALF) and lung biopsies when the patient is scheduled for routine bronchoscopies in the follow-up period.

This study involves measurements of EBP and PFR done by the particles in exhaled air (PExA) system on lung transplanted patients with and without acute or chronic rejection. The patients who do not develop any form of rejection will serve as a control group to the ones who develop rejection. Furthermore, each patient will serve as their own control.

The purpose of this study is to find better means of identifying rejection of transplanted lungs in earlier stages, and to explore candidate biomarkers. Earlier diagnosis of rejection of the transplanted organ can lead to better treatment possibilities and a positive impact on survival after LTx.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone LTx at Skåne University Hospital, SUS Lund

Exclusion Criteria:

* None

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing lung transplantation at Skåne University Hospital, SUS Lund.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-09-18 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Concentration of proteins in EBP | Pre-transplantation
  Proteins from exhaled air are collected onto a membrane for subsequently molecular analysis. Analysis aims to identify candidate biomarker for acute and chronic rejection of transplanted lungs.
Concentration of proteins in EBP | Day 1-3 after lung transplantation
  Proteins from exhaled air are collected onto a membrane for subsequently molecular analysis. Analysis aims to identify candidate biomarker for acute and chronic rejection of transplanted lungs.
Concentration of proteins in EBP | 1 month after lung transplantation
  Proteins from exhaled air are collected onto a membrane for subsequently molecular analysis. Analysis aims to identify candidate biomarker for acute and chronic rejection of transplanted lungs.
Concentration of proteins in EBP | 3 months after lung transplantation
  Proteins from exhaled air are collected onto a membrane for subsequently molecular analysis. Analysis aims to identify candidate biomarker for acute and chronic rejection of transplanted lungs.
Concentration of proteins in EBP | 6 months after lung transplantation
  Proteins from exhaled air are collected onto a membrane for subsequently molecular analysis. Analysis aims to identify candidate biomarker for acute and chronic rejection of transplanted lungs.
Concentration of proteins in EBP | 9 months after lung transplantation
  Proteins from exhaled air are collected onto a membrane for subsequently molecular analysis. Analysis aims to identify candidate biomarker for acute and chronic rejection of transplanted lungs.
Concentration of proteins in EBP | 12 months after lung transplantation
  Proteins from exhaled air are collected onto a membrane for subsequently molecular analysis. Analysis aims to identify candidate biomarker for acute and chronic rejection of transplanted lungs.
Concentration of proteins in EBP | 18 months after lung transplantation
  Proteins from exhaled air are collected onto a membrane for subsequently molecular analysis. Analysis aims to identify candidate biomarker for acute and chronic rejection of transplanted lungs.
Concentration of proteins in EBP | 2 years after lung transplantation
  Proteins from exhaled air are collected onto a membrane for subsequently molecular analysis. Analysis aims to identify candidate biomarker for acute and chronic rejection of transplanted lungs.
Concentration of proteins in EBP | 3 years after lung transplantation
  Proteins from exhaled air are collected onto a membrane for subsequently molecular analysis. Analysis aims to identify candidate biomarker for acute and chronic rejection of transplanted lungs.
Concentration of proteins in EBP | 4 years after lung transplantation
  Proteins from exhaled air are collected onto a membrane for subsequently molecular analysis. Analysis aims to identify candidate biomarker for acute and chronic rejection of transplanted lungs.
Particle flow rate from the airways (PFR) | Day 1-3 after transplantation
  PFR will be measured by the PExA device. The flow rate and the particle pattern will be analysed to find differences between groups of lung transplanted patients with and without rejection.
Particle flow rate from the airways (PFR) | 1 month after transplantation
  PFR will be measured by the PExA device. The flow rate and the particle pattern will be analysed to find differences between groups of lung transplanted patients with and without rejection.
Particle flow rate from the airways (PFR) | 3 months after transplantation
  PFR will be measured by the PExA device. The flow rate and the particle pattern will be analysed to find differences between groups of lung transplanted patients with and without rejection.
Particle flow rate from the airways (PFR) | 6 months after transplantation
  PFR will be measured by the PExA device. The flow rate and the particle pattern will be analysed to find differences between groups of lung transplanted patients with and without rejection.
Particle flow rate from the airways (PFR) | 9 months after transplantation
  PFR will be measured by the PExA device. The flow rate and the particle pattern will be analysed to find differences between groups of lung transplanted patients with and without rejection.
Particle flow rate from the airways (PFR) | 12 months after transplantation
  PFR will be measured by the PExA device. The flow rate and the particle pattern will be analysed to find differences between groups of lung transplanted patients with and without rejection.
Particle flow rate from the airways (PFR) | 18 months after transplantation
  PFR will be measured by the PExA device. The flow rate and the particle pattern will be analysed to find differences between groups of lung transplanted patients with and without rejection.
Particle flow rate from the airways (PFR) | 2 years after transplantation
  PFR will be measured by the PExA device. The flow rate and the particle pattern will be analysed to find differences between groups of lung transplanted patients with and without rejection.
Particle flow rate from the airways (PFR) | 3 years after transplantation
  PFR will be measured by the PExA device. The flow rate and the particle pattern will be analysed to find differences between groups of lung transplanted patients with and without rejection.
Particle flow rate from the airways (PFR) | 4 years after transplantation
  PFR will be measured by the PExA device. The flow rate and the particle pattern will be analysed to find differences between groups of lung transplanted patients with and without rejection.

SECONDARY OUTCOMES:
Concentration of proteins and other biomarkers in plasma | Pre-transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in plasma
Concentration of proteins and other biomarkers in plasma | Day 1 after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in plasma
Concentration of proteins and other biomarkers in plasma | Day 2 after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in plasma
Concentration of proteins and other biomarkers in plasma | Day 3 after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in plasma
Concentration of proteins and other biomarkers in plasma | 1 month after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in plasma
Concentration of proteins and other biomarkers in plasma | 3 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in plasma
Concentration of proteins and other biomarkers in plasma | 6 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in plasma
Concentration of proteins and other biomarkers in plasma | 9 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in plasma
Concentration of proteins and other biomarkers in plasma | 12 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in plasma
Concentration of proteins and other biomarkers in plasma | 18 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in plasma
Concentration of proteins and other biomarkers in plasma | 2 years after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in plasma
Concentration of proteins and other biomarkers in plasma | 3 years after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in plasma
Concentration of proteins and other biomarkers in plasma | 4 years after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in plasma
Concentration of proteins and other biomarkers in BAL | Day 1-3 after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in BAL
Concentration of proteins and other biomarkers in BAL | 1 month after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in BAL
Concentration of proteins and other biomarkers in BAL | 3 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in BAL
Concentration of proteins and other biomarkers in BAL | 6 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in BAL
Concentration of proteins and other biomarkers in BAL | 9 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in BAL
Concentration of proteins and other biomarkers in BAL | 12 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in BAL
Concentration of proteins and other biomarkers in BAL | 18 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in BAL
Concentration of proteins and other biomarkers in BAL | 2 years after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in BAL
Concentration of proteins and other biomarkers in BAL | 3 years after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in BAL
Concentration of proteins and other biomarkers in BAL | 4 years after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in BAL
Concentration of proteins and other biomarkers in lung tissue | At the time of lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in lung tissue. Both taken from the native lung and from the donor lung.
Concentration of proteins and other biomarkers in lung tissue | 1 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in lung tissue
Concentration of proteins and other biomarkers in lung tissue | 3 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in lung tissue
Concentration of proteins and other biomarkers in lung tissue | 6 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in lung tissue
Concentration of proteins and other biomarkers in lung tissue | 9 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in lung tissue
Concentration of proteins and other biomarkers in lung tissue | 12 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in lung tissue
Concentration of proteins and other biomarkers in lung tissue | 18 months after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in lung tissue
Concentration of proteins and other biomarkers in lung tissue | 2 years after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in lung tissue
Concentration of proteins and other biomarkers in lung tissue | 3 years after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in lung tissue
Concentration of proteins and other biomarkers in lung tissue | 4 years after lung transplantation
  Concentration and composition of proteins and other biomarkers will be analysed in lung tissue

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Lindstedt, MD, PhD, Principal Investigator — Region Skåne, Lund University
Locations (1):
- Skåne University Hospital, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ericson PA, Mirgorodskaya E, Hammar OS, Viklund EA, Almstrand AR, Larsson PJ, Riise GC, Olin AC. Low Levels of Exhaled Surfactant Protein A Associated With BOS After Lung Transplantation. Transplant Direct. 2016 Aug 26;2(9):e103. doi: 10.1097/TXD.0000000000000615. eCollection 2016 Sep. PMID 27795995
- [Background] Stenlo M, Hyllen S, Silva IAN, Bolukbas DA, Pierre L, Hallgren O, Wagner DE, Lindstedt S. Increased particle flow rate from airways precedes clinical signs of ARDS in a porcine model of LPS-induced acute lung injury. Am J Physiol Lung Cell Mol Physiol. 2020 Mar 1;318(3):L510-L517. doi: 10.1152/ajplung.00524.2019. Epub 2020 Jan 29. PMID 31994907
- [Background] Broberg E, Hyllen S, Algotsson L, Wagner DE, Lindstedt S. Particle Flow Profiles From the Airways Measured by PExA Differ in Lung Transplant Recipients Who Develop Primary Graft Dysfunction. Exp Clin Transplant. 2019 Dec;17(6):803-812. doi: 10.6002/ect.2019.0187. Epub 2019 Oct 11. PMID 31615381
- [Background] Behndig AF, Mirgorodskaya E, Blomberg A, Olin AC. Surfactant Protein A in particles in exhaled air (PExA), bronchial lavage and bronchial wash - a methodological comparison. Respir Res. 2019 Sep 26;20(1):214. doi: 10.1186/s12931-019-1172-1. PMID 31558154